CLINICAL TRIAL: NCT00265486
Title: Erythropoietin Protect the Cerebral Blood Flow and Oxygenation During Simulated Dive?
Brief Title: Can Erythropoietin Protect the Cerebral Blood Flow and Oxygenation During Simulated Dive?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Kjeld, 1. reservelæge, Rigshospitalet, Denmark
Other Study IDs: KF 01 271889
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2005-08

CONDITIONS: Healthy
Keywords: Divers; Brain; Flow; Blood; EPO; Dive; reflex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Recombinant human Erythropoietin — Adm 100 U/kg sc 1 hour before completing exercise in protocol

SUMMARY:
During facial cooling and especially during breath hold, can mammals - and also humans - elicit a so called dive reflex, causing bradycardia, peripheral vasoconstriction and centralization of blood flow to brain, lungs and heart but the reflex is suppressed by physical activity. The dive reflex can be elicited by breath hold alone and will be more pronounced during simultaneously facial cooling, but not by stimulation of other skin receptors.

The dive reflex has an oxygen conserving effect, because of intense vasoconstriction in both viscera and muscles, and simultaneously with reduction in cardiac output (CO). Therefore plasma lactate will rise, to compensate for the lesser regional blood flow. If one hyperventilates with 100 % oxygen, then the reflex can still be elicited, but it is more pronounced during asphyxia. Experienced sports divers, who has been diving for more than 7-10 years have reduced post apnea acidosis and oxidational stress, but probably also less sensitivity for progressive hypoxia and hypercapnia, because these individuals have a more pronounced dive reflex.

Transcranial Doppler ultrasonography (TCD) gives a reproducibly value for brain perfusion by continuously non-invasive real-time sampling. A single piezo-electrical transducer sends and collects ultrasound through the temporal region of the scull, where it is the thinnest. Hereby can the blood flow of arteria cerebri anterior, media (MCA) and posterior and basilaris be estimated.

With TCD it can be shown that the cerebral blood flow rises in MCA in healthy subjects during facial cooling, with normal ventilation, when resting in a supine position without affecting the systemic blood pressure. Single Photon Emission Computerized Tomography (SPECT)-scanning during normo-baric and hyperbaric pressure of professional divers breathing 100 % oxygen has shown to reduce the cerebral blood flow in several regions of the brain.

But it is yet unknown how brain blood flow and metabolism are affected by an "face immersion dive" and simultaneously prolonged physical activity, and hence a rise in lactate under hyperbaric pressure (3 meters), breathing atmospheric air, similar to the circumstances for trained scuba divers work.

Presumably it will cause a fall in brain blood flow and in time cognitive deficits.

Erythropoietin (rhEPO) is a well known drug, used as doping in sports for about 15 years. So far the only known enhancement in athletic achievement by rhEPO is caused by peripheral improvements and especially blood capability to transport oxygen to the working muscles; this has been documented by a rise in haematocrit. rhEPO has also a neuroprotective effect on neurons in patients with neuron damage caused by cerebral hypoxic ischeamia.

rhEPO work also on a series of cerebral mechanisms, including enhanced motor and spatial learning and more. Enhanced motor learning may improve the professional divers choices during work and may be also physical performance and mechanical efficiency. Intravenous injection of rhEPO will increase rhEPO in cerebrospinal fluids, since rhEPO is capable of crossing blood brain. All together this may indicate that rhEPO, not only works on physical performance, but also has effects on the brain. rhEPO has also an effect on the condition of cancer and dialysis patients, not only explained by merely increased hematocrit.

This project will add new knowledge in the understanding of the mechanisms of clinical use of rhEPO.

The purpose of this study is to investigate, how brain blood flow and metabolism are affected by face immersion dive and simultaneously breath hold during normo-baric and hyperbaric pressure (3 m depth) when breathing atmospheric air in trained sports divers. IL-6, HSP-72, lactate, ammonium and body-temperature will be measured. Brain and muscle oxygenation will be measured by near-infrared spectroscopi (NIRS). Furthermore we will investigate whether a small dose of rhEPO affects mentioned parameters during simulated dive in pressure chamber with facial cooling.

Hypothesis Brain blood flow in trained divers will be diminished during prolonged physical activity during simultaneously face immersion dive and breath hold under hyperbaric pressure.

There will be a release of IL-6 and HSP-72. Pretreatment with a small amount of rhEPO before prolonged physical activity during simulated dive has a protective effect on brain blood flow and oxygenation.

DETAILED DESCRIPTION:
Background

During facial cooling and especially during breath hold, can mammals - and also humans - elicit a so called dive reflex, causing bradycardia, peripheral vasoconstriction and centralization of blood flow to brain, lungs and heart (18 Foster et al 2005), but the reflex is suppressed by physical activity. The dive reflex can be elicited by breath hold alone and will be more pronounced during simultaneously facial cooling, but not by stimulation of other skin receptors (19 Asmussen et al 1968).

Intrapleural pressure and lung volume affects the dive reflex in a way so that the less part of vital capacity being used, the more pronounced bradycardia. This is explained by the fact that the pulmonary stretch receptors are activated less by smaller lung volumes and thereby sending a smaller vagal afferent output.

The dive reflex has an oxygen conserving effect, because of intense vasoconstriction in both viscera and muscles, and simultaneously with reduction in cardiac output (CO). Therefore plasma lactate will rise, to compensate for the lesser regional blood flow. If one hyperventilates with 100 % oxygen, then the reflex can still be elicited, but it is more pronounced during asphyxia. Experienced sports divers, who has been diving for more than 7-10 years have reduced post apnea acidosis and oxidational stress (18 Foster et al 2005), but probably also less sensitivity for progressive hypoxia and hypercapnia, because these individuals have a more pronounced dive reflex.

Persons with sleep apnea are, like trained breath hold divers, exposed for repetitive episodes of hypoxia and hypercapnia during their sleep, of up to 30 to 60 seconds, and they have developed a lesser sensitivity for this. These patients does typically have chronically higher activity of the sympathetic nervous system, higher peripheral resistance and blood pressure (18 Foster et al 2005).

SCUBA Sports divers, who dive more than 100 times a year, especially in cold water have diminished cerebral blood flow and a cognitive deficit (20 Slosman et al 2003). Age and body mass index (BMI) are associated to diminished cerebral blood flow and the cognitive deficit, possibly because, SCUBA divers with higher BMI, have larger pools of nitrogen in their adipose tissues, which then gives smaller non-symptomatic incidences of decompression sickness (20 Slosman et al 2003). But is obvious to assume, that it could be caused by diminished cerebral blood flow, because of the dive reflex.

Also climbing to high altitudes (between 54488 and 8848 m) is shown to give cognitive deficit. Those who had the most pronounced symptoms, where very sensitive to hypoxia by hyperventilation. It was suspected, that hypocapnia because of hyperventilation was causing diminished cerebral blood flow (33 Hornbein TF et al 1989).

Transcranial Doppler ultrasonography (TCD) gives a reproducibly value for brain perfusion by continuous non-invasive real-time sampling (14 Aslid et al 1982). A single piezo-electrical transducer sends and collects ultrasound through the temporal region of the scull, where it is the thinnest. Hereby can the blood flow of arteria cerebri anterior, media (MCA) and posterior and basilaris be estimated.

With TCD it can be shown which parts of the brain, that are activated during static and dynamic work (15 Colebatch et al 1991, 16 Dahl et al 1992). Also vasodilatation when CO2 is high is seen as a rise in arterial blood flow, and small emboli sends a characteristic signal during carotid surgery (17 Halsey et al 1986).

With Blood Oxygenation Level-Dependent functional Magnetic Resonance imaging, BOLD fMRI is it shown that breath hold induced hypercapnia gives a higher cerebral blood flow in sensorimotor cortex, frontal cortex, in ganglia basale, in visual cortex and in cerebellum (21 Kastrup et al 1999). The largest changes are seen in cerebellum and the smallest in frontal cortex (21 Kastrup et al 1999).

With TCD it can be shown that the cerebral blood flow rises in MCA in healthy subjects during facial cooling, with normal ventilation, when resting in a supine position without affecting the systemic blood pressure (22 Browna et al 2003). Single Photon Emission Computerized Tomography (SPECT)-scanning during normo-baric and hyperbaric pressure of professional divers breathing 100% oxygen has shown to reduce the cerebral blood flow in several regions of the brain (23 Di Pieroa et al 2002).

The brain metabolism depends on a continuously supply of glucose, which is suppressed during the hypoglycemia induced by prolonged work (1 Nybo et al 2003). The brain is though capable of using other substrates to a certain extent , like lactate which is absorbed in an amount proportionally with the arterial concentration (2 Dalsgaard et al 2003). So it seems that the brain during prolonged work is capable of having an absorption of lactate to the same amount as glucose. Also it seems that lactate is being metabolized, since it is not accumulated in spinal fluid or brain tissue (3 Madsen et al 1999). At rest the brain absorption of glucose is balanced by a proportional oxygen absorption (approximately 1:6). When the brain is activated, this equilibrium is disturbed regionally (4 Fox Raichle et al 1986) and globally (5 Madsen 1995). At rest, where the concentration of lactate in serum is low, is the importance of lactate for brain metabolism minimal, but during physical activity, where plasma lactate rises, is the absorption increasing and it contributes to the lowering in brain metabolic ratio.

The underlying cause for the fall in brain metabolic ratio during physical activity is not known. But the excessive amount of carbohydrate (in proportion to oxygen ) can reach a level, comparable to the total amount of brain glycogen (6 Dalsgaard et al 2004).

Also the activated brain seems to free IL-6 and HSP-72 (7 Nybo et al 2002). On the other hand only a small amount of ammonium is absorbed by the brain (8 Nybo et al 2005), which partly - besides a rise in temperature (9 Nybo et al 2002) - explains, why brain autoregulation is less stable during especially intense physical activity (10 Ogoh et al 2005), as known from patients in coma caused by hepatic failure (11 Larsen et al 1996).

A possible explanation for the fall in brain metabolic ratio during physical activity is that this mechanism can be overruled in rat brain after administration of the non-specific beta-blocking drug propanolol (12 Schmalbruch et al 2002), while the cardioselective drug metoprolol does not have the same effect in humans (13 Dalsgaard et al 2004).

But it is yet unknown how brain blood flow and metabolism are affected by an "face immersion dive" and simultaneously prolonged physical activity, and hence a rise in lactate under hyperbaric pressure (3 m dybde), breathing atmospheric air, similar to the circumstances for trained scuba divers work.

Presumably it will cause a fall in brain blood flow and in time cognitive deficits.

Erythropoietin (rhEPO) is a well known drug, used as doping in sports for about 15 years (24 Parisotto R et al, 2001). So far the only known enhancement in athletic achievement by rhEPO is caused by peripheral improvements and especially blood capability to transport oxygen to the working muscles (25 A Gaudard et al, 2003); this has been documented by a rise in haematocrit (25 A Gaudard et al, 2003). rhEPO has also a neuroprotective effect on neurones in patients with neuron damage caused by cerebral hypoxic ischeamia (26, HH Marti 2004).

rhEPO work also on a series of cerebral mechanisms, including enhanced motor and spatial learning, increased dopamine production and improved neural function through activation of calcium-channels (26, HH Marti 2004). Enhanced motor learning may improve the professional divers choices during work and may be also physical performance and mechanical efficiency. Less dopamine-concentration in the brain can cause enhanced fatigue, and increased dopamine production caused by treatment with rhEPO may delay fatigue during physical activity. Intravenous injection of rhEPO will increase rhEPO in cerebrospinal fluids, since rhEPO is capable of crossing blood brain (26, HH Marti 2004). All together this may indicate that rhEPO, not only works on physical performance, but also has effects on the brain. An enhanced concentration of rhEPO could improve brain function by stimulating neural function and thereby induce increased release of dopamine, reduce mismatch between oxygen and glucose absorption, improve voluntarily activation and increase effect through improved motor learning. rhEPO has also an effect on the condition of cancer and dialysis patients, not only explained by merely increased heamocrit (27, W Jelkmann, 2004).

This project will add new knowledge in the understanding of the mechanisms of clinical use of rhEPO.

Erythropoietin (EPO) is a heamatopoietic growth factor primarily synthesized in the kidneys. It stimulates erythropoiesis. New investigations has shown that EPO can be neuroprotective in cerebral ischaemia, brain trauma, autoimmune encephalomyelitis and kainattoksicitet (26, HH Marti 2004)). The pathophysiology is yet unknown, but may secondarily to gene induction, through suppression of the inflammatory response, such as inducible nitrogen oxide synthesis (iNOS) and mitogen activated protein kinase (MAPK), to suppress apoptosis. Also it may be plausible, that EPO upregulates antioxidants. In rats rhEPO has increased survival after circulatory shock, induced by total ischemia / reperfusion of the splanchnicus (28 F Squadrito et al, 1999). Treatment with rhEPO suppressed activity of endotoxin mediated increase in NO. rhEPO suppresses the production of iNOS in smooth muscle cells after stimulation of the proinflammatory IL-1. These effects of rhEPO are expressed from hours to days after treatment with rather high solitary doses and seems to be independently mediated by the erythropoietic effect, which can only be achieved after weeks continuous treatment with rhEPO (29 E Kusano et al, 1999, 30 Brines ML et al, 2000).

Purpose of this study The purpose of this study is to investigate, how brain blood flow and metabolism are affected by face immersion dive and simultaneously breath hold during normo-baric and hyperbaric pressure (3 m depth) when breathing atmospheric air in trained sports divers. IL-6, HSP-72, lactate, ammonium and body-temperature will be measured. Brain and muscle oxygenation will be measured by near-infrared spectroscopi (NIRS). Furthermore we will investigate whether a small dose of rhEPO affects mentioned parameters during simulated dive in pressure chamber with facial cooling.

Hypothesis Brain blood flow in trained divers will be diminished during prolonged physical activity during simultaneously face immersion dive and breath hold under hyperbaric pressure when breathing atmospheric air.

There will be a release of IL-6 and HSP-72. Pretreatment with a small amount of rhEPO before prolonged physical activity during simulated dive has a protective effect on brain blood flow and oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* No smokers
* Healthy, including no history of cardiopulmonary disease
* Normal heart and lung stethoscopy
* Active diving at least twice a week
* V02max at least 15 METS
* Signed and informed consent

Exclusion Criteria:

* Smokers
* Any condition needing drug treatment

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 12 healthy non-smoking free divers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2005-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kjeld, MD, Principal Investigator — Rigshospitalet, dept of aneasthesiolgy, 2042, Blegdamsvej, 2100 CPH, DK
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen East, Denmark

REFERENCES:
- [Background] Brines ML, Ghezzi P, Keenan S, Agnello D, de Lanerolle NC, Cerami C, Itri LM, Cerami A. Erythropoietin crosses the blood-brain barrier to protect against experimental brain injury. Proc Natl Acad Sci U S A. 2000 Sep 12;97(19):10526-31. doi: 10.1073/pnas.97.19.10526. PMID 10984541
- [Background] Squadrito F, Altavilla D, Squadrito G, Campo GM, Arlotta M, Quartarone C, Saitta A, Caputi AP. Recombinant human erythropoietin inhibits iNOS activity and reverts vascular dysfunction in splanchnic artery occlusion shock. Br J Pharmacol. 1999 May;127(2):482-8. doi: 10.1038/sj.bjp.0702521. PMID 10385249
- [Background] Parisotto R, Wu M, Ashenden MJ, Emslie KR, Gore CJ, Howe C, Kazlauskas R, Sharpe K, Trout GJ, Xie M. Detection of recombinant human erythropoietin abuse in athletes utilizing markers of altered erythropoiesis. Haematologica. 2001 Feb;86(2):128-37. PMID 11224480
- [Background] Di Piero V, Cappagli M, Pastena L, Faralli F, Mainardi G, Di Stani F, Bruti G, Coli A, Lenzi GL, Gagliardi R. Cerebral effects of hyperbaric oxygen breathing: a CBF SPECT study on professional divers. Eur J Neurol. 2002 Jul;9(4):419-21. doi: 10.1046/j.1468-1331.2002.00436.x. PMID 12099928
- [Background] Brown CM, Sanya EO, Hilz MJ. Effect of cold face stimulation on cerebral blood flow in humans. Brain Res Bull. 2003 Jun 30;61(1):81-6. doi: 10.1016/s0361-9230(03)00065-0. PMID 12788210
- [Background] Kastrup A, Kruger G, Glover GH, Neumann-Haefelin T, Moseley ME. Regional variability of cerebral blood oxygenation response to hypercapnia. Neuroimage. 1999 Dec;10(6):675-81. doi: 10.1006/nimg.1999.0505. PMID 10600413
- [Background] Slosman DO, De Ribaupierre S, Chicherio C, Ludwig C, Montandon ML, Allaoua M, Genton L, Pichard C, Grousset A, Mayer E, Annoni JM, De Ribaupierre A. Negative neurofunctional effects of frequency, depth and environment in recreational scuba diving: the Geneva "memory dive" study. Br J Sports Med. 2004 Apr;38(2):108-14. doi: 10.1136/bjsm.2002.003434. PMID 15039241